CLINICAL TRIAL: NCT01432678
Title: Vitamin D Status in Pediatric Asthma
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Orathai Piboonpocanun, Department of Pediatrics, Faculty of Medicine, Siriraj Hospital, Mahidol University
Other Study IDs: 744/2553(EC1)
Record Dates: First submitted 2011-09-10; First posted 2011-09-13 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D; asthma
MeSH Terms: conditions — Vitamin D Deficiency; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- asthma patients: controlled asthma partly controlled asthma uncontrolled asthma

SUMMARY:
The purpose of this study is to evaluate level of vitamin D in pediatric asthma and relationship between vitamin D and level control of asthma.

DETAILED DESCRIPTION:
cross-sectional study

ELIGIBILITY:
Inclusion Criteria:

* children between the age of 6 years and 18 years with the diagnosis of asthma who are attending the outpatient pediatric department, pediatric allergy clinic

Exclusion Criteria:

* patients who have chronic pulmonary, heart disease, chronic renal failure, liver disease, endrocrine disorder, or receieve antiepileptic drugs, vitamin D supplement

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: allergy clinic in tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Orathai Piboonpocanun, Principal Investigator — Siriraj Hospital
Locations (1):
- Division of Allergy and Immunology, Department of Pediatrics, Faculty of medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Result] Krobtrakulchai W, Praikanahok J, Visitsunthorn N, Vichyanond P, Manonukul K, Pratumvinit B, Jirapongsananuruk O. The effect of vitamin d status on pediatric asthma at a university hospital, Thailand. Allergy Asthma Immunol Res. 2013 Sep;5(5):289-94. doi: 10.4168/aair.2013.5.5.289. Epub 2013 Aug 12. PMID 24003385